CLINICAL TRIAL: NCT00003157
Title: A Phase I Study of Gemcitabine, Cisplatin, and Radiation Therapy in Patients With Locally Advanced Pancreatic and Gastric Cancer
Brief Title: Radiation Therapy and Chemotherapy in Treating Patients With Cancer of the Pancreas or Stomach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-964352; CDR0000065949 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-30 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Cisplatin; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiation + gemcitabine + cisplatin (Experimental): Patients undergo radiotherapy to the tumor and lymph nodes, followed by a decrease in radiotherapy to the tumor alone. Radiation therapy is administered for a total of 5.5 weeks. Patients receive intravenous gemcitabine twice weekly over the first 3 weeks of radiotherapy. Cisplatin is administered intravenously twice weekly following gemcitabine therapy. Three patients are treated at each dose level. Dose escalation does not occur until all patients at a given dose level have completed radiotherapy and returned for a 4 week follow up. Patients exhibiting stable disease remain on therapy until disease progression or intolerable toxic effects. Patients experiencing toxic effects and no disease progression are retreated at a lower dose. Patients are followed every 3 months for the first 2 years then every 6 months for the next year.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of radiation therapy plus chemotherapy in treating patients who have cancer of the pancreas or stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of gemcitabine and cisplatin that can be administered during a standard course of radiation therapy for patients with unresectable or locally recurrent pancreatic and gastric cancer. II. Describe the tolerance of gemcitabine, cisplatin, and radiation therapy in this patient population. III. Seek preliminary evidence of the therapeutic activity of this regimen in this patient population as measured by survival.

OUTLINE: This is a dose escalation study. Patients undergo radiotherapy to the tumor and lymph nodes, followed by a decrease in radiotherapy to the tumor alone. Radiation therapy is administered for a total of 5.5 weeks. Patients receive intravenous gemcitabine twice weekly on Tuesday and Friday over the first 3 weeks of radiotherapy. Cisplatin is administered intravenously twice weekly following gemcitabine therapy. Three patients are treated at each dose level. Dose escalation does not occur until all patients at a given dose level have completed radiotherapy and returned for a 4 week follow up. The dose limiting toxicity (DLT) is defined as the dose at which at least 2 of 6 patients experience unacceptable toxic effects. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences DLT. Patients exhibiting stable disease remain on therapy until disease progression or intolerable toxic effects. Patients experiencing toxic effects and no disease progression are retreated at a lower dose. Patients are followed every 3 months for the first 2 years then every 6 months for the next year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unresectable (including incomplete resections) or locally recurrent pancreatic or gastric cancer No evidence of metastases outside of the planned radiation field No cystadenocarcinoma of the pancreas or pancreatic tumors of neuroendocrine origin

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-1 Life Expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin within normal limits Alkaline phosphatase no greater than 3.0 times upper limit of normal (ULN) AST no greater than 3.0 times ULN Renal: Creatinine no greater than 1.3 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception No significant infection or medical illness No significant nausea or vomiting At least 1200 calories per day of oral nutrition

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent biologic therapy Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy (except focal fields for skin cancer that do not overlap with planned radiotherapy fields) Surgery: At least 21 days since laparotomy surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1998-02; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 3 years

SECONDARY OUTCOMES:
Survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James A. Martenson, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Martenson JA Jr, Viglitotti AG, Geeraerts LH, et al.: Phase I study of twice weekly gemcitabine (GEM) and cisplatin (CDDP) during radiation therapy (RT) for advanced pancreas and gastric cancer: a progress report. [Abstract] Proceedings of the American Society of Clinical Oncology A-2305, 2001.